CLINICAL TRIAL: NCT06835959
Title: Development of a Mobile Health Intervention to Improve Blood Pressure Management in Pregnancy (Moms@Home)
Brief Title: Moms@Home: A Storytelling-based Mobile Health Intervention to Improve Blood Pressure Management in Pregnancy
Acronym: Moms@Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lara Kovell, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00001895; K23HL163450 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Hypertension in Pregnancy; Chronic Hypertension; Gestational Hypertension
Keywords: Hypertension in pregnancy; Moms@Home; Mobile health intervention; Blood pressure; Blood pressure management; Hypertension; Gestational hypertension; Storytelling; Home blood pressure monitoring; Storytelling mobile intervention
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either the Moms@Home intervention or ESC through permuted blocked randomization, in blocks of multiples of 2 such that half of the participants will use Moms@Home and the other half ESC.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the randomization assignments. Both investigators and participants will be aware of the randomization assignments to facilitate the implementation of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moms@Home arm (Experimental): Participants randomized to Moms@Home will receive the Moms@Home app (± Samsung smartphone) to self-report data including home blood pressure monitoring values from a digital blood pressure monitor and physical activity data from a FitBit activity tracker.
  Interventions: Behavioral: Moms@Home
- Enhanced Standard Care arm (Active Comparator): Participants randomized to Enhanced Standard Care (ESC) will receive a paper diary to self-report data including measurements from a digital blood pressure monitor.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Moms@Home — Participants will use a storytelling mobile health app for daily home-based blood pressure monitoring and symptom/medication adherence tracking.
  Other Names: Peer Support Intervention
  Arms: Moms@Home arm
Behavioral: Enhanced Standard of Care — Participants will use a paper journal daily to track home-based blood pressure values
  Other Names: Self-tracking Journal
  Arms: Enhanced Standard Care arm

SUMMARY:
This pilot study will examine the effects of a digital health approach, Moms@Home, on home blood pressure monitoring in a diverse population of pregnant women with hypertension.

DETAILED DESCRIPTION:
The study aims to standardize and test a storytelling approach to promote HBPM and improve BP management and pregnancy-specific outcomes in pregnant women with Hypertension (HTN). The study will integrate three components to improve BP care and outcomes: 1) the Moms@Home mobile app to promote HBPM through storytelling videos and a patient dashboard of BP data, 2) a digital BP monitor for HBPM, and 3) an HBPM report that curates and shares key health data with the right provider at the right time. Designed by and for pregnant women with HTN across racial/ethnic groups, the Moms@Home intervention is novel because it leverages digital health, behavior change techniques, and culturally relevant storytelling to improve HTN self-care while facilitating patient/caregiver communication through an HBPM report. Investigators are conducting a pilot randomized controlled trial (RCT) of Moms@Home vs. enhanced standard care, with plans to enroll 100 pregnant women (50% from racial/ethnic minority groups) with gestational or chronic HTN to determine whether Moms@Home vs. enhanced standard care (BP monitor, diary) improves HBPM adherence (primary outcome) and to evaluate the feasibility, acceptability, and sustainability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* English or Spanish speaking
* A diagnosis of gestational (20-26 weeks gestational age) or chronic hypertension (8-26 weeks gestational age)
* Singleton or multiple gestation pregnancy,
* A patient of the University of Massachusetts Memorial Health Obstetrics/Maternal and Fetal Medicine clinics in Worcester, Massachusetts
* Willing to share home blood pressure monitoring data
* Comfortable with the use of smartphones and mobile apps

Exclusion Criteria:

* Severe hypertension (Systolic blood pressure ≥160 mmHg or Diastolic blood pressure ≥100 mmHg)
* Current diagnosis of preeclampsia
* Active substance use
* Serious physical illness (e.g., unable to interact with a smart device)
* Enrolled in another home blood pressure monitoring program
* Excluded from study participation by their provider
* Inability to provide informed consent
* Prisoners/institutionalized individuals

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-11-16 (Estimated)

PRIMARY OUTCOMES:
Home Blood Pressure Monitoring Adherence | 8 weeks
  Home blood pressure monitoring (HBPM) adherence is defined as performing HBPM measures ≥3 out of 7 days/week
Feasibility of the Moms@Home intervention | 8 weeks
  Among the participants in the intervention group, the feasibility of the Moms@Home intervention will be assessed through a post-intervention survey using a 5-point Likert scale, with questions on the value and overall satisfaction with the mobile intervention app. On a numeric scale, number of screened and eligible participants and the number/reason(s) for declining participation or withdrawal will be tracked.
Acceptability | 8 weeks
  Acceptability will be assessed using the System Usability Scale (SUS) and the perceived impact section of the End-user Mobile Application Rating Scale (uMARS). These are both validated measures of the usability/quality of mobile health apps. SUS is scored on a 0-100 scale, a higher score meaning better usability. The uMARS is scored on a 5-point Likert scale, with the total score calculated by averaging the scores across the items within the perceived impact subscale.

SECONDARY OUTCOMES:
Self-Efficacy | Baseline, 4 weeks, 8 weeks
  Change in self-efficacy will be determined through the Self-Efficacy to Manage Hypertension scale (Warren-Findlow, 2012). Each item of this scale is scored on a 1 to 10 scale, with the total score calculated by averaging the scores across the items. Higher mean scores indicate higher self-efficacy.
Sustainability | 8 weeks
  The sustainability of the Moms@Home intervention will be assessed through a post-intervention survey using a 5-point Likert scale, evaluating participants' perceptions of whether the Moms@Home storytelling mobile app could be continued beyond the study period.
Blood Pressure (BP) measures | Baseline, 4 weeks, 8 weeks
  Home Blood Pressure Monitoring (HBPM) values will be assessed using blood pressure data collected from the Moms@Home app and paper BP diaries. Clinic blood pressure values will be obtained through a review of electronic health records.
Engagement with Moms@Home | 4 weeks, 8 weeks
  Among the participants in the intervention group, engagement with the Moms@Home intervention will be measured on a numeric scale by number of logins, time spent in the app, surveys completed, and storytelling videos watched.
Medication Adherence | Baseline, 4 weeks, 8 weeks
  On a numeric scale, baseline and change in medication adherence will be assessed through a baseline, midpoint and post-intervention survey.
Medication titration | Baseline, 4 weeks, 8 weeks
  Medication titration will be assessed based on any changes in the blood pressure medications participants are taking. These changes may include adjustments in dosage, discontinuation of medications, initiation of new medications, or switching between different medications. This data will be obtained from participants' electronic health records.
Goal attainment | Baseline, 8 weeks
  Attainment of personal goals related to home blood pressure monitoring set at the study baseline will be assessed with a post-intervention survey and reported as a percentage of goal achieved.
Physical Activity | Baseline, 4 weeks, 8 weeks
  On numeric scale, baseline and change in physical activity will be tracked by daily steps recorded by the FitBit.

OTHER OUTCOMES:
Focus group interviews | At least 3 months after randomization
  The investigators will perform qualitative focus groups in a subpopulation of the Moms@Home study assignment to assess for ease of use, barriers and facilitators related to the intervention and long-term maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Kovell, MD,MSc, Principal Investigator — University of Massachusetts Medical School, Worcester
Locations (1):
- UMass Memorial Medical Center - Memorial Campus, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will consist of de-identified self-reported demographic and behavioral data from participants, along with home blood pressure monitoring (HBPM) data and physical activity data from the Moms@Home app and FitBit device. We will work with the NHLBI BioData Catalyst (BDC) to deposit the appropriate data. Otherwise, this final dataset will be kept on hand and distributed upon reasonable request after an appropriate data-use agreement has been put in place. All data will be de-identified prior to release.
Supporting Information: ICF
Time Frame: November 23rd, 2027 - November 23rd, 2028
Access Criteria: The NHLBI Other investigators with appropriate data use agreements

REFERENCES:
- [Background] McManus DD, Trinquart L, Benjamin EJ, Manders ES, Fusco K, Jung LS, Spartano NL, Kheterpal V, Nowak C, Sardana M, Murabito JM. Design and Preliminary Findings From a New Electronic Cohort Embedded in the Framingham Heart Study. J Med Internet Res. 2019 Mar 1;21(3):e12143. doi: 10.2196/12143. PMID 30821691
- [Background] Hirshberg A, Sammel MD, Srinivas SK. Text message remote monitoring reduced racial disparities in postpartum blood pressure ascertainment. Am J Obstet Gynecol. 2019 Sep;221(3):283-285. doi: 10.1016/j.ajog.2019.05.011. Epub 2019 May 20. No abstract available. PMID 31121137
- [Background] Pealing LM, Tucker KL, Mackillop LH, Crawford C, Wilson H, Nickless A, Temple E, Chappell LC, McManus RJ; OPTIMUM-BP Investigators. A randomised controlled trial of blood pressure self-monitoring in the management of hypertensive pregnancy. OPTIMUM-BP: A feasibility trial. Pregnancy Hypertens. 2019 Oct;18:141-149. doi: 10.1016/j.preghy.2019.09.018. Epub 2019 Oct 13. PMID 31618706
- [Background] Dodson JA, Schoenthaler A, Fonceva A, Gutierrez Y, Shimbo D, Banco D, Maidman S, Olkhina E, Hanley K, Lee C, Levy NK, Adhikari S. Study design of BETTER-BP: Behavioral economics trial to enhance regulation of blood pressure. Int J Cardiol Cardiovasc Risk Prev. 2022 Oct 31;15:200156. doi: 10.1016/j.ijcrp.2022.200156. eCollection 2022 Dec. PMID 36573193
- [Background] Schoenthaler A, Cruz J, Payano L, Rosado M, Labbe K, Johnson C, Gonzalez J, Patxot M, Patel S, Leven E, Mann D. Investigation of a Mobile Health Texting Tool for Embedding Patient-Reported Data Into Diabetes Management (i-Matter): Development and Usability Study. JMIR Form Res. 2020 Aug 31;4(8):e18554. doi: 10.2196/18554. PMID 32865505
- [Background] Warren-Findlow J, Seymour RB, Brunner Huber LR. The association between self-efficacy and hypertension self-care activities among African American adults. J Community Health. 2012 Feb;37(1):15-24. doi: 10.1007/s10900-011-9410-6. PMID 21547409
- [Background] Aquino M, Munce S, Griffith J, Pakosh M, Munnery M, Seto E. Exploring the Use of Telemonitoring for Patients at High Risk for Hypertensive Disorders of Pregnancy in the Antepartum and Postpartum Periods: Scoping Review. JMIR Mhealth Uhealth. 2020 Apr 17;8(4):e15095. doi: 10.2196/15095. PMID 32301744
- [Background] Jakubowski BE, Hinton L, Khaira J, Roberts N, McManus RJ, Tucker KL. Is self-management a burden? What are the experiences of women self-managing chronic conditions during pregnancy? A systematic review. BMJ Open. 2022 Mar 18;12(3):e051962. doi: 10.1136/bmjopen-2021-051962. PMID 35304393
- [Background] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800
- [Background] Kovell LC, Denu M, Revoori R, Sadaniantz K, Staples B, Chiriboga G, Forrester SN, Lemon SC, Moore Simas TA, Person S, McManus DD, Mazor KM. Barriers and facilitators to home blood pressure monitoring in women with pregnancies complicated by hypertensive disorders: a qualitative study. J Hypertens. 2024 Nov 1;42(11):1994-2002. doi: 10.1097/HJH.0000000000003835. Epub 2024 Aug 9. PMID 39248134
- Available data/document: Informed Consent Form: Informed consent form — https://drive.google.com/file/d/1q09u34SVFOO2TXC7vXuDAE0MAjJfgVyA/view?usp=drive_link

DOCUMENTS (2):
  • Study Protocol (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT06835959/Prot_000.pdf
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT06835959/ICF_001.pdf